CLINICAL TRIAL: NCT01977430
Title: Randomized Open Clinical Trial to Compare the Effectiveness of the Administration of Diuretics in Hemodialysis Patients With Residual Renal Function in Single Centre
Brief Title: Clinical Trial to Compare Effectiveness of Diuretics in Hemodialysis Patients With Residual Renal Function
Acronym: RRF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Maria Isabel Bolós Contador, Medica Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEF-DIU-2013-CSPT; CSPT2013/058 (Other: Ethics Committee Corporació Sanitària Parc Taulí)
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Kidney Insufficiency; Hemodialysis Treatment; Diuresis Preserved
Keywords: Residual renal function; Combined thiazide-furosemide therapy; Haemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Hydrochlorothiazide; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diuretics arm (Experimental): The diuretic arm's patients will receive combined thiazide-furosemide therapy for 1 month: 20 mg of furosemide three times daily and 50 mg of hydrochlorothiazide twice daily
  Interventions: Drug: Hydrochlorothiazide and furosemide
- Control Arm (No Intervention)

INTERVENTIONS:
Drug: Hydrochlorothiazide and furosemide — This clinical trial is cross-over study. The diuretic arm's patients will receive combined diuretic treatment for 1 month: 20 mg of furosemide three times daily and 50 mg of hydrochlorothiazide twice daily
  Arms: Diuretics arm

SUMMARY:
Introduction: Chronic kidney disease is characterized by a progressive deterioration of renal function. At the end of the progression, when complications occur (overhydration, electrolyte imbalances or retention of uremic toxins), a percentage of patients requiring renal replacement therapy (haemodialysis). When starting the haemodialysis, the patient holds the residual renal function (RRF) which is lost over time. To preserve the RRF, the patient is treated with diuretics loops and / or thiazide diuretics. The effect of this treatment is lost when renal function worsens. In this context, there are few studies that explore the use and effectiveness of diuretics in patients on haemodialysis 2. Objectives and Hypothesis:

Hypothesis: The treatment with furosemide and hydrochlorothiazide in haemodialysis patients with RRF could:

* To decrease in weight gain between haemodialysis sessions.
* To increase urine volume.
* To decrease the ultrafiltration in haemodialysis sessions ( the long interdialytic interval)

Main Objective:To asses the effect of combined hydrochlorothiazide-furosemide therapy on gain weight between haemodialysis sessions in patients with RRF

Secondary Objective: To asses the effect of combined hydrochlorothiazide-furosemide therapy on dialytic, clinical and analytical variables and use of the antihypertensive treatment

3. Methodology: Randomized open clinical trial to compare the effectiveness of the administration of diuretics in haemodialysis patients with residual renal function in single centre.

The population of study are patients with chronic renal disease in haemodialysis therapy that they preserve residual renal function ( more 200ml daily of urine). It will be a simple randomization, to asses the effect of combined hydrochlorothiazide-furosemide therapy

After a of 15 days washout without diuretic treatment, patients will be randomized to receive or not receive combined diuretic treatment for 1 month. After a 1 month washout , the patients will be receive or not the treatment according to cross over trial.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Chronic kidney disease, stage 5 Chronic Kidney Disease, in haemodialysis
* Renal residual function preserved(more or equal 200 ml daily of urine)
* Minimum 3 months on haemodialysis and wish to participate in this study

Exclusion criteria:

* Less 4 millequivalent of potassium plasma in interdialytic sessions or to require potassium intradialytic treatment.
* Less 1 Kg of gain weight in the long interdialytic interval.
* Adverse effects with treatment in the past.
* To refusal to participate in the study.
* Pregnancy or lactation period.
* Contraindication the use of diuretic therapy, according to pharmacological profile.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
To asses the effect of combined hydrochlorothiazide-furosemide therapy on weight gain between haemodialysis sessions in patients with RRF | 14 weeks
  Gain weight

SECONDARY OUTCOMES:
To asses the effect of combined hydrochlorothiazide-furosemide therapy on dialytic, clinical and analytical variables and use of the antihypertensive treatment | 14 weeks
  Variations of the next parameters in the different periods(15 days, 1, 2 and 3 months) of the clinical trial:
  urine volume, reduction of ultrafiltration in interdialysis sessions and long interdialytic interval, dry weight, blood pressure intradialysis,plasma potassium, plasma bicarbonate, plasma uric acid, urinary sodium, urinary chloro and urinary potassium in interdialytic sessions . Use of the antihypertensive treatment. To Appear complications for example: hypotensions, cramps and symptomatic hyperuricemia. Creatinine clearance and urea clearance. Use of potassium treatment intradialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mabel - Bolos-Contador, MD, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain